CLINICAL TRIAL: NCT06584188
Title: The Effect of Anti-inflammatory Cryoagent on the Level of Postoperative Pain in Patients with Symptomatic Irreversible Pulpitis and Apical Periodontitis.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, abdulrahman ziad elwadiah, abdelrahman_ziad_kasem@dent.asu.edu.eg, Ain Shams University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DentAinShams
Record Dates: First submitted 2024-02-11; First posted 2024-09-04 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intra-radicular saline at room temperature (Experimental): * Final flush with 20 mL of saline solution
  * At room temperature for 5 minutes.
  * Three samples will be collected from periapical fluid .
  Interventions: Drug: anti-inflammatory ketorolac tromethamine

INTERVENTIONS:
Drug: anti-inflammatory ketorolac tromethamine — * Intra- radicular anti-inflammatory {ketorolac tromethamine at room temperature}.
  * Intra- radicular cold anti-inflammatory {ketorolac tromethamine at 2-5C}.

SUMMARY:
* The aim of this study is comparative between:

  1. Intra-radicular cryotherapy using cold anti-inflammatory {ketorolac tromethamine at 2-5C}.
  2. Intra-radicular final flush anti-inflammatory {ketorolac tromethamine at room temperature}.
* In terms of:

C. Level of post-operative pain {POP} using a visual analog scale {VAS}. D. Level of substance P in periapical fluid will be analyzed by enzyme-linked immunosorbent assay (ELISA) kit.

Outcomes :

* Primary outcomes: Level of Post-operative pain.
* Secondary outcomes: Level of substance P expression

ELIGIBILITY:
Inclusion Criteria:

1. Patients that will be diagnosed with symptomatic irreversible pulpitis and apical periodontitis.
2. Patient age ranging from 18-40 years.
3. Males or females.
4. Lower premolars.
5. Medically free patients.
6. Teeth with mature apex.
7. Teeth without any type of root resorption.

Exclusion Criteria:

1. Patients with other pulpal diagnosis.
2. Medically compromised patients.
3. Vulnerable group; pregnant females, mentally ill, etc...
4. Patients taking analgesics or anti-inflammatory drugs.
5. Teeth with open apex.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Level of Post-operative pain. | 12 hours post operative
  measure intensity of post operative pain using visual analogue scale that was represented by a 100 mm horizontal ruler with no number markings other than a 0 at one end and a 10 at the other end. The following categories of postoperative pain levels were used to assess pain: 0 indicating no pain, mild pain (1-3), moderate pain (4-7) and severe pain (8-10)
Level of Post-operative pain. | 24 hours post operative
  measure intensity of post operative pain using visual analogue scale that was represented by a 100 mm horizontal ruler with no number markings other than a 0 at one end and a 10 at the other end. The following categories of postoperative pain levels were used to assess pain: 0 indicating no pain, mild pain (1-3), moderate pain (4-7) and severe pain (8-10)
Level of Post-operative pain. | 48 hours post operative
  measure intensity of post operative pain using visual analogue scale that was represented by a 100 mm horizontal ruler with no number markings other than a 0 at one end and a 10 at the other end. The following categories of postoperative pain levels were used to assess pain: 0 indicating no pain, mild pain (1-3), moderate pain (4-7) and severe pain (8-10)

SECONDARY OUTCOMES:
Level of substance P expression. | 15 minutes following access cavity preparation.
  Quantification of substance P will be done using an ELISA test from peri-radicular fluid swab.
Level of substance P expression. | 30 minutes following access cavity preparation.
  Quantification of substance P will be done using an ELISA test from peri-radicular fluid swab.
Level of substance P expression. | Immediately prior to obturation
  Quantification of substance P will be done using an ELISA test from peri-radicular fluid swab.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided